CLINICAL TRIAL: NCT02685319
Title: Mapping Human Muscle Satellite Cell Fate By Real-Time
Brief Title: Mapping Human Muscle Satellite Cell Fate By Real-Time Imaging
Acronym: S48
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1512016862
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Flaccid Muscle Tone
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- muscle biopsy (Experimental): a muscle sample will be taken from the mid-thigh (Vastus Lateralis) and analyzed
  Interventions: Procedure: muscle biopsy

INTERVENTIONS:
Procedure: muscle biopsy — a muscle sample will be taken from the mid-thigh (Vastus Lateralis) and analyzed

SUMMARY:
Mapping Human Muscle Satellite Cell Fate By Real-Time Imaging

DETAILED DESCRIPTION:
The aim of this study is to obtain human muscle samples for cell culturing to analyze muscle cell development in real-time to uncover factors that influence growth.

ELIGIBILITY:
-Inclusion Criteria:

* men 20-29 yrs
* BMI between 20 and 34.9
* Fasting Glucose <110 mg/dL
* Blood Pressure <160/100mm Hg
* Non-Diabetic
* LDL-Cholesterol <160mg/dL
* Triacylglycerol <400 mg/dL
* Makers of kidney, liver, and heart functions within 10% of clinical normalcy
* <1.5hr /wk of habitual aerobic exercise training and no resistance exercise training in the past 6 months

Exclusion Criteria:

* men <20or>29 yrs

  * BMI between <20 and >34.9
  * Fasting Glucose >110 mg/dL
  * Blood Pressure >160/100mm Hg
  * Non-Diabetic
  * LDL-Cholesterol >160mg/dL
  * Triacylglycerol >400 mg/dL
  * Pre-existing kidney or liver conditions

    -->1.5hr /wk of habitual aerobic exercise training and no resistance exercise training in the past 6 months
  * Currently taking prescribed blood thinners

Ages: 20 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mapping Human Muscle Satellite Cell Fate By Real-Time Imaging | <10 hrs
  this study is to obtain human muscle samples for cell culturing which will be exposed to a novel real-time imaging technique in order to elucidate factors that influence muscle satellite cell growth.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University - Stone Hall 700 W State St, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No